CLINICAL TRIAL: NCT01498159
Title: Health Promoters and Pharmacists in Diabetes Team Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ben Gerber, Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-0099; R01DK091347 (NIH)
Record Dates: First submitted 2011-12-15; First posted 2011-12-23 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Pharmacists; Community Health Aides
MeSH Terms: conditions — Diabetes Mellitus | interventions — Physicians, Primary Care; Electronic Health Records; Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist + Health Promoter (Experimental): Participants in this group will receive support from both a pharmacist and health promoter. Number of sessions will be determined by the study team member and patient.
  Interventions: Behavioral: Pharmacist disease/medication management; Behavioral: Pharmacist-patient encounters; Behavioral: Pharmacist medication intensification and adherence support; Behavioral: Pharmacist communication with primary care physicians; Behavioral: Pharmacist documentation in electronic medical record; Behavioral: Health promoter-patient encounters in-person or by phone; Behavioral: Health promoter medication and lifestyle support; Behavioral: Health promoter communication with pharmacists
- Pharmacist (Active Comparator): Participants will receive support from pharmacist.
  Interventions: Behavioral: Pharmacist disease/medication management; Behavioral: Pharmacist-patient encounters; Behavioral: Pharmacist medication intensification and adherence support; Behavioral: Pharmacist communication with primary care physicians; Behavioral: Pharmacist documentation in electronic medical record

INTERVENTIONS:
Behavioral: Pharmacist disease/medication management
Behavioral: Pharmacist-patient encounters
Behavioral: Pharmacist medication intensification and adherence support
Behavioral: Pharmacist communication with primary care physicians
Behavioral: Pharmacist documentation in electronic medical record
Behavioral: Health promoter-patient encounters in-person or by phone
  Arms: Pharmacist + Health Promoter
Behavioral: Health promoter medication and lifestyle support
  Arms: Pharmacist + Health Promoter
Behavioral: Health promoter communication with pharmacists
  Arms: Pharmacist + Health Promoter

SUMMARY:
This research evaluates a diabetes management intervention designed to improve medication adherence and intensify therapy to reach goals in blood sugar, blood pressure, and cholesterol levels. This study will determine the benefit and cost of adding community health promoters to pharmacist disease management services. If there is benefit, then this approach may help reduce the burden of diabetes and its related complications among minorities with diabetes.

DETAILED DESCRIPTION:
Many African-Americans and Latinos with diabetes do not achieve the recommended goals for normal blood sugar, blood pressure, or cholesterol level, placing them at high risk for complications. This study will evaluate the impact of a novel intervention designed to improve lifestyle behaviors and medication adherence, and intensify therapy to reach goals. The first component of the intervention includes a clinic-based pharmacist disease management program. The program includes detailed patient assessments, physician-approved treatment plans, patient education and support services to enhance medication adherence. In addition, this program includes intensification of medication therapy to improve blood sugar, blood pressure, and cholesterol levels to reach recommended goals. The second component of the intervention includes health promoters (HPs), or community-based lay health workers. Health promoters are commonly found in minority communities and provide assistance for individuals overcoming language, cultural, and other barriers to conventional health care services. They may provide autonomy support and solve problems related to medication adherence barriers. Furthermore, health promoters may complement pharmacist activities by improving access to medications, assisting in continuity of care with providers, monitoring response to therapy, and reinforcing educational messages. The proposed study will determine whether the addition of health promoters to clinic based pharmacist service delivery improves care. The study will involve the recruitment of 300 African-American and Latino adults with uncontrolled diabetes through the University of Illinois Medical Center in Chicago and randomization to one of two groups: (1) pharmacist management (Pharm) for 12 months; or (2) pharmacist management with HP support (Pharm+HP) for 12 months. Cross-over will occur at 12 months such that the Pharm group will be intensified by the addition of HP support and HP support will be phased out from the Pharm+HP group to assess maintenance. The specific aims include: (1) To evaluate the effectiveness of Pharm+HP compared with Pharm alone on diabetes behaviors (including healthy eating, physical activity, and medication adherence), hemoglobin A1c, blood pressure, and LDL-cholesterol levels; (2) To evaluate the maintenance of improved diabetes behaviors as well as clinical outcomes by phasing out HP support from the Pharm+HP group after year 1; (3) To evaluate the intensification offered by adding an HP after one year of Pharm alone; and (4) To evaluate the cost and cost-effectiveness of Pharm+HP and Pharm alone.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Latino/Hispanic or African-American
* Verbal fluency in English or Spanish
* Age 21 or above
* History of type 2 diabetes (> 1 year)
* Hemoglobin A1c ≥ 8.0% (within 1 year)
* Receives primary care at UIMC (> 1 year)
* Taking at least one oral medication for diabetes or hypertension

Exclusion Criteria:

* Unable to verbalize comprehension of study or impaired decision making (e.g., dementia)
* Lives outside Chicago communities of recruitment (3+ months/year)
* Household member already participating in same study
* Plans to move from the Chicago area within the next year
* Pregnant or trying to get pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-12; Primary Completion 2016-04 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 24 months
  Hemoglobin A1c

SECONDARY OUTCOMES:
Diabetes Knowledge | 24 months
  Diabetes Knowledge
Autonomous Self-Regulation | 24 months
  Autonomous Self-Regulation
Perceived Competence | 24 months
  Perceived Competence
Medication Adherence | 24 months
  Medication Adherence
Body mass index | 24 months
  Body mass index
Diabetes Self-Care Behaviors | 24 months
  Diabetes Self-Care Behaviors
Quality of Life | 24 months
  Quality of Life
Healthcare Utilization | 24 months
  Healthcare Utilization
Systolic Blood Pressure | 24 months
  Systolic Blood Pressure
Diastolic Blood Pressure | 24 months
  Diastolic Blood Pressure
LDL Cholesterol | 24 months
  LDL Cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Ben S Gerber, MD, MPH, Principal Investigator — University of Illinois at Chicago; Lisa K Sharp, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Gerber BS, Cano AI, Caceres ML, Smith DE, Wilken LA, Michaud JB, Ruggiero LA, Sharp LK. A pharmacist and health promoter team to improve medication adherence among Latinos with diabetes. Ann Pharmacother. 2010 Jan;44(1):70-9. doi: 10.1345/aph.1M389. Epub 2009 Dec 22. PMID 20028957
- [Background] Gerber BS, Rapacki L, Castillo A, Tilton J, Touchette DR, Mihailescu D, Berbaum ML, Sharp LK. Design of a trial to evaluate the impact of clinical pharmacists and community health promoters working with African-Americans and Latinos with diabetes. BMC Public Health. 2012 Oct 23;12:891. doi: 10.1186/1471-2458-12-891. PMID 23088168
- [Result] Sharp LK, Tilton JJ, Touchette DR, Xia Y, Mihailescu D, Berbaum ML, Gerber BS. Community Health Workers Supporting Clinical Pharmacists in Diabetes Management: A Randomized Controlled Trial. Pharmacotherapy. 2018 Jan;38(1):58-68. doi: 10.1002/phar.2058. Epub 2017 Nov 30. PMID 29121408
- [Derived] Nabulsi NA, Yan CH, Tilton JJ, Gerber BS, Sharp LK. Clinical pharmacists in diabetes management: What do minority patients with uncontrolled diabetes have to say? J Am Pharm Assoc (2003). 2020 Sep-Oct;60(5):708-715. doi: 10.1016/j.japh.2020.01.024. Epub 2020 Feb 27. PMID 32115392
- [Derived] Locatelli SM, Sharp LK, Syed ST, Bhansari S, Gerber BS. Measuring Health-related Transportation Barriers in Urban Settings. J Appl Meas. 2017;18(2):178-193. PMID 28961153
- See also: IHRP Study Description — http://www.ihrp.uic.edu/study/health-promoters-and-pharmacists-diabetes-team-management